CLINICAL TRIAL: NCT04916353
Title: Effects of Ultrasound-guide Hypertonic Dextrose Injection for Chronic Subacromial Bursitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, ShihWei Huang, Attending Physician, Taipei Medical University Shuang Ho Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N201812061
Record Dates: First submitted 2021-06-02; First posted 2021-06-07 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Chronic Shoulder Pain
Keywords: Prolotherapy; subacromial bursitis; ultrasound
MeSH Terms: interventions — Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 20% hypertonic dextrose water injection group (Experimental): echo guide 20% dextrose water 3ml was injection in lesion site
  Interventions: Drug: hypertonic dextrose water
- Steroid injection group (Active Comparator): Triamcinolone Acetonide 40mg/ml, 1ml, and Lidocaine 2ml as the active comparator group
  Interventions: Drug: Triamcinolone Acetonide.

INTERVENTIONS:
Drug: hypertonic dextrose water — 20% hypertonic dextrose water injection for chronic shoulder pain
  Other Names: Prolotherapy group
  Arms: 20% hypertonic dextrose water injection group
Drug: Triamcinolone Acetonide. — Triamcinolone Acetonide 40mg/1ml injection
  Other Names: comparatice group
  Arms: Steroid injection group

SUMMARY:
The aim of this study is to investigate the echoguide hypertonic injection and compared steroid injection in subacromial bursitis patients about clinical and ultrasound image presentation.

DETAILED DESCRIPTION:
Subacromial bursitis is one of the major causes of chronic refractory shoulder pain. It can cause patients with shoulder pain when shoulder exercise and heavy lifting and limiting the range of motion. It can also influence the sleep quality due to pain symptoms of the shoulder. Usually, these patients had limited response to medication and physical modality. Steroid injection was often adopted for intervention, but the adverse effects should be considered. Therefore, prolotherapy was taken as an alternative treatment for chronic subacromial bursitis. It involves the injection of small volumes of an irritant agent, most commonly a hyperosmolar dextrose solution, at the lesion site. Hyperosmolar dextrose appears to be the most commonly used agent today. The aim of this study is to investigate hypertonic injections in subacromial bursitis patients about clinical and ultrasound image presentation. The investigators conducted a double-blinded randomized controlled trial for 60 participants with chronic shoulder pain for 3 months with subacromial bursitis. In the study group, the echo guide 20% dextrose water was injected into the lesion site, and the control group received the echo guide steroid injection. ROM, SPADI, VAS, x-ray, and ultrasound data were obtained at baseline. At weeks 2, 6, 12, ROM, SPADI, VAS, and ultrasound data were evaluated. The ANOVA and independent t-test are applied for analysis by SPSS 20.0 with a P value less than 0.05 as statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Aged more than 20 years old with diagnosis of chronic supraspinatus tendinosis by ultrasound and clinical shoulder pain lasting for more than 3 months.

Exclusion Criteria:

* History of shoulder fracture and operation, with frozen shoulder or full thickness ruptur of rotator cuff, steroid, or hyaluronic acid, or platelet rich plasma (PRP) injection during the period of intervention and following up.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Shoulder Pain and Disability Index (change of SPADI) | Week0 Week2 Week6 Week12
  Shoulder Pain and Disability Index (SPADI), a self-administered assessment tool that was used to measure pain and disability related to shoulder disease. The SPADI consists of 5 pain and 8 disability items that are measured on a visual analog scale. Pain and disability subscales were calculated as the mean of the corresponding items on a 0-100 scale; the highest score indicated the most severe pain and disability. The total outcome score used for statistical analysis was calculated as the sum of the pain and disability subscales.

SECONDARY OUTCOMES:
Ultrasound | Week0 Week2 Week6 Week12
  The ultrasound evaluated the thickness of subarcomial bursa
Shoulder ROM (Range of Motion) | Week0 Week2 Week6 Week12
  Pain-free passive range of motion (PROM) of the shoulder was designated as the range of motion attained at the most painful position and was measured using a digital goniometer in 6 directions flexion, extension, abduction, adduction, external rotation and internal rotation. Five directions of the shoulder joint were measured (flexion, abduction, adduction, internal rotation, and external rotation) while participants were lying in a supine position. Additionally, shoulder extension was measured in the side-lying position.
Pain (VAS, Visual Analogue Scale) | Week0 Week2 Week6 Week12
  Shoulder pain was assessed according to an 11-point numerical rating scale (NRS). This tool was simple to use and was highly correlated with the visual analog scale, verbal rating scale, and Faces Pain Scale-Revised. The NRS is considered a valid and reliable pain assessment tool. The pain intensity was graded from 0 (no pain) to 10 (the most intense level of pain). The participants reported their pain level at rest and during the movement of shoulder joint in all direction. The most painful movement score was used for further data analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Lien-Chieh Lin, Study Chair — Taipei Medical University-Shuang Ho Hospital,Ministry of Health and Welfare
Locations (2):
- Taiwan (2):
  - Shuang Ho Hospital, New Taipei City, Zhonghe Dist
  - Taipei Medical University-Shuang Ho Hospital,Ministry of Health and Welfare, New Taipei City, Zhonghe Dist

IPD SHARING:
Plan to Share IPD: No